CLINICAL TRIAL: NCT04059718
Title: SCI Thrive: Efficacy of a Peer-led Online Self-Management Program
Acronym: SCIThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor Department of Rehabilitation Medicine University of Washington School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006621
Record Dates: First submitted 2019-08-12; First posted 2019-08-16 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment arm will be enrolled in the SCI Thrive Peer-Led Online Self-Management program and will take part in the next available group session.
  Interventions: Behavioral: SCI Thrive Peer-Led Online Self-Management Program
- Wait-list Control (No Intervention): Wait-list control arm will only complete assessments during the 6 week group period. Subjects will be offered a place in the SCI Thrive Peer-Led Online Self-Management program after 6 weeks and completing the assessments.

INTERVENTIONS:
Behavioral: SCI Thrive Peer-Led Online Self-Management Program — 6 week online course in self-management for individuals with spinal cord injuries. This was developed by a team using principles of cognitive behavioral techniques.
  Arms: Treatment

SUMMARY:
SCI Thrive is a randomized controlled trial to test the efficacy of SCI Thrive (6 week Peer-Led Online Self-Management Program) to improve quality of life and self-efficacy for individuals with SCI.

DETAILED DESCRIPTION:
With spinal cord injury (SCI), individuals are at a greater risk for a number of chronic health conditions. Research suggests that these health conditions reduce quality of life for individuals with SCI and decrease social engagement. Many of these health conditions are in fact preventable by early detection, behavioral changes, and early intervention.

Self-management programs have emerged as an adjunct to traditional health care services based management of chronic conditions. Self-management programs provide necessary knowledge, and skills, but ultimately focus on the central role of the individual in balancing medical management, maintaining life roles and community engagement, and managing emotional distress.

Beyond self-management strategies alone, more evidence now exists for increasing self-management and knowledge of health related resources for individuals with SCI through peer support. Face-to-face peer support programs have been found to improve self-efficacy and reduce the occurrence of medical complications. Additionally, peer support is positively associated with social participation and life satisfaction.

The purpose of this study is to determine if an online, peer led self-management program can lead to:

1. An improvement in of quality of life for people with spinal cord injuries
2. Increase in confidence in your ability to achieve goals (self-efficacy) and community participation
3. Assess if improvements last 3 months after completion
4. Evaluate participant satisfaction with the program and the materials

If you decide to take part in this study, you will first be asked to complete an online survey which should take about 20 minutes. You will then be randomized (like flipping a coin) in the treatment group or the control group. If you are in the treatment group, you will begin the online program. If you are in the control group, you will be asked to wait 6 weeks before beginning the program. After 6 weeks, both groups will take a second online survey. If you are in the control group, we will ask if you want to take part in the online program. If you do, you will have one additional survey upon completion of the online program. 3 months after completion of the online program, we will contact you to complete the final online survey. Each of these surveys should take approximately 15 minutes.

The first survey will ask some information about you and your background. The first survey and the last two will also ask questions about how you manage your health with a spinal cord injury, how satisfied you are in various aspects of your life, how much you get around, how you spend your time, and interact with people. Some of the most sensitive questions ask about satisfaction with income, relationships, and sexual activity. You may refuse to answer any question in the surveys.

When you take part in the online self-management program, you will work through a different educational module each week. These will include modules on goal setting, thinking strategies and distraction, alternative thoughts, problem solving and decision tools, communication and advocacy, applying to your own goals, and relaxations exercises for each session. Each module should take approximately 1 hour to complete.

During the 6 week program, there will be at lease three video/telephone conferences with the peer leader and the other participants. The goal of the weekly conference is for participants to discuss the materials, what aspects are working or not working for them, provide their individual perspectives, and support each other. These conferences will last no longer than 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Online: Any Location
* Spinal Cord Injury
* Age >= 18 years
* English Speaking
* Cognitively able to engage in the course and able to complete initial start-up requirements on the course website
* Computer/Smartphone/Tablet with internet access

Exclusion Criteria:

* Planned absence during the 6 week course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Quality of Life Scale (PQOL) | Collected at enrollment, 6 weeks, and 3 months post treatment
  The PQOL measures satisfaction with 12 different aspects of life including an individual's contact with family or friends, contribution to the community, meaning and purpose in life, and happiness.
Change in Self-Efficacy for Managing Chronic Disease 6-item Scale (SMCD) | Collected at enrollment, 6 weeks, and 3 months post treatment
  Self-Efficacy for Managing Chronic Disease 6-item Scale (SMCD) is a measure of self-efficacy for managing chronic disease in core domains of symptom control, role function, emotional functioning, and communicating with physicians. It has been found to be reliable and valid and has been translated into other languages.
Change in Life Space Assessment (LSA) | Collected at enrollment, 6 weeks, and 3 months post treatment
  Life Space Assessment (LSA) is a self-report measure that captures the extent and frequency of environmental mobility (life space) and participation of persons with mobility limitations. It includes assessment of the need for personal assistance and/or equipment. It has been found to be a reliable and valid measure in persons with SCI.
Change in the Craig Handicap Assessment and Reporting Technique (CHART) Short Form | Collected at enrollment, 6 weeks, and 3 months post treatment
  The CHART is a reliable and valid assessment of participation and has been used frequently with individuals with SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- Northwest Regional Spinal Cord Injury System: University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.